CLINICAL TRIAL: NCT00825292
Title: Detection and Classification of Colon Polyps: A Comparison of High Definition White Light and Narrow Band Imaging (Endoscopic Trimodal Imaging; ETMI)
Brief Title: Detection and Classification of Colon Polyps
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Seth A. Gross, M.D. and Michael B. Wallace, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-002653 00
Record Dates: First submitted 2007-12-26; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Colon Polyps
Keywords: colon polyps, colon adenomas
MeSH Terms: conditions — Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): HDNBI colonoscopy followed by standard white light colonoscopy
  Interventions: Procedure: Polp removal and identification; Procedure: ETMI colonoscope (ETMI scope is a FDA approved device)
- 1 (Active Comparator): standard white light colonoscopy followed by HDNBI colonoscopy
  Interventions: Procedure: colon polyp removal; Procedure: ETMI colonoscope (ETMI scope is a FDA approved device)

INTERVENTIONS:
Procedure: Polp removal and identification — Identify polyp during colonoscopy then remove polyp
  Other Names: Colonoscopy with polypectomy
  Arms: 2
Procedure: colon polyp removal — identify and remove polyp
  Other Names: Colonoscopy with polypectomy
  Arms: 1
Procedure: ETMI colonoscope (ETMI scope is a FDA approved device) — ETMI colonoscope used to identify colon polyps as compared to HD white light colonoscope identifying colon polyps.
  Other Names: Detecting and removing colon polyps

SUMMARY:
Colon cancer is the third most common cancer in western society. To prevent colon cancer it is recommended for people to undergo a screening colonoscopy at the age of fifty. The purpose of the colonoscopy is to remove polyps, since some of these lesions are precancerous. Precancerous polyps are called adenomas. This method of prevention is effective, but the standard colonoscopy currently used does not detect all polyps. Studies have reported a polyp miss rate of about 24%. Furthermore, we are unable to distinguish precancerous polyps from benign polyps, also known as hyperplastic polyps, with standard colonoscopy. This results in all polyps being removed at time of colonoscopy, even the benign polyps.

To help improve the detection of colon polyps new endoscopic technologies have been developed. These technologies include high definition white light (HDWL)and high definition narrow band imaging (HDNBI). HDWL improves the overall resolution of the images seen during colonoscopy. HDNBI can help us better classify polyps by enhancing their tissue appearance as well as seeing small blood vessels and capillaries.

The goal of this study to determine if HDNBI imaging shows an increased polyp detection rate when compared to the current standard colonoscopy. In addition to develop a classification system to help better differentiate between precancerous polyps and their benign counterparts using HDWL and HDNBI.

DETAILED DESCRIPTION:
II. Hypothesis:

1. The use of NBI colonoscopy will reduce the miss rate for colon polyps compared to standard white light imaging.
2. HDWl and HDNBI are more accurate than standard colonoscopy for the classification of adenomatous polyps in comparison to other non-premalignant polyps.

III. Specific Aims:

1. Compare the miss rate of standard white light imaging compared to NBI for detection of colon polyps with NBI
2. Estimate the accuracy of standard white light, HDWL and HDNBI imaging modes for the classification of adenomatous (premalignant) versus non-adenomatous (hyperplastic, inflammatory, normal) polyps.
3. Examine the inter-observer agreement for classification of adenomatous versus non-adenomatous polyps based on standard, NBI and HDWL imaging.

IV. Research Design and Methods:

4.1 Study Design: A prospective phase II cross-over trial. Patients will undergo both procedures (standard, NBI) back to back under conscious sedation. The order of the procedure will be randomized.

4.2 Setting: The study will take place at Mayo Clinic Jacksonville, Division of Gastroenterology, an expert center in the diagnosis and treatment of colon polyps.

4.3 Study Subjects All patients scheduled for colonoscopy at Mayo Clinic Jacksonville will be screened for eligibility using inclusion and exclusion criteria. The patients that are deemed eligible will be offered participation in the study. Informed consent will be obtained and the participant will be registered in our database. Prior to consent the participant will be made aware of the investigative nature of the study, alternatives, risks, and benefits.

4.4 Eligibility Criteria

Inclusion Criteria:

1. Age 18 years or older.
2. Informed written consent.

Exclusion Criteria:

1. History of inflammatory bowel disease.
2. Patients with severe cardiopulmonary disease precluding colonoscopy.
3. Presence of conditions not allowing for polypectomy or biopsy (e.g. coagulation disorder).
4. Known familial polyposis syndrome (FAP, HNPCC, Juvenile polyposis, etc)
5. Sub-optimal preparation for the procedure, which will be determined by patient history or based on the initial colonoscopy.
6. Pregnancy

4.5 Procedure and Data Collections

A. Pre-procedure:

All patients will be prepared for colonoscopy with the standard preparation and will be scheduled to have the procedure at Mayo Clinic Jacksonville. The principal investigator (PI) will screen eligible patients based on medical history, physical exam and laboratory data on day of procedure.

Patients typically arrive at the registration area at least 60 minutes before start of scheduled procedure. A GI endoscopy nurse will prepare patients in the standard manner and intravenous access will be placed. Eligible patients will be offered informed consent by the study PI or designee. Patients who agree to participate in the study will sign informed consent and will be registered in the database. A log with only non-identifiable (e.g. patients # 1) will also be maintained of eligible patients who decline to participate. The GI endoscopy nurse will monitor patient's vitals before, during and after procedure as per standard protocol.

B. Procedure:

The exams will be performed back to back with a standard colonoscope and an ETMI colonoscope provided by Olympus. The order of the first and second procedure will be randomized according to a list prepared by the statistician using randomly permuted blocks to ensure equal numbers of patients are randomized to the two groups. All patients will be sedated with meperidine or fentanyl and midazolam to achieve conscious sedation. Each procedure will be preformed by a different endoscopist. The endoscopist will be either the P.I. supervised by a GI staff physician or solely by one of the five GI staff physicians. During the initial colonoscopy all visualized polyps will be noted, photographed, and removed. When the ETMI colonoscope is used, all polyps will be photographed using these modes (HDWL, HDNBI). The NBI portion of the exam will be performed using the MB-046 cap to further enhance stabilization of the focal length of the colonoscope.

The second procedure will be done with the same level of careful inspection as the first although we not specifically regiment the time of withdrawal beyond what the endoscopist feels is necessary for a careful examination. During the second colonoscopy all visualized polyps will be noted, photographed and removed. During the first procedure, the time will be evaluated with a stopwatch. The stopwatch will start when the endoscopist begins pull-back at the cecum and end when the scope is removed from the anal verge. The clock will be stopped during washing of the bowel, polypectomy, biopsy or any other therapeutic maneuver. At the end of the first procedure, the endoscopist will be informed of the withdrawal and inspection time and every effort will be made to match this to the second procedure. Time will be recorded similarly for the second procedure. Polyps will be classified as pedunculated, raised-sessile (rounded) or flat. Flat polyps will be further classified according to the Paris endoscopic classification 14.

C. Post-procedure:

After the procedure all patients will be brought to the recovery and monitored as per standard protocol. Participants will be given discharge instructions as per protocol and also be provided with information to contact the P.I. if any problems should occur. Any post procedure complication will be reviewed on weekly intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Informed written consent

Exclusion Criteria:

1. History of inflammatory bowel disease.
2. Patients with severe cardiopulmonary disease precluding colonoscopy.
3. Presence of conditions not allowing for polypectomy or biopsy (e.g. coagulation disorder).
4. Known familial polyposis syndrome (FAP, HNPCC, Juvenile polyposis, etc)
5. Sub-optimal preparation for the procedure, which will be determined by patient history or based on the initial colonoscopy.
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
1. Compare the miss rate of standard white light imaging compared to NBI for detection of colon polyps with NBI | 2 years

SECONDARY OUTCOMES:
2. Estimate the accuracy of standard white light, HDWL and HDNBI imaging modes for the classification of adenomatous (premalignant) versus non-adenomatous (hyperplastic, inflammatory, normal) polyps. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Seth A. Gross, M.D., Principal Investigator — Mayo Clinic; Michael B. Wallace, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Jemal A, Tiwari RC, Murray T, Ghafoor A, Samuels A, Ward E, Feuer EJ, Thun MJ; American Cancer Society. Cancer statistics, 2004. CA Cancer J Clin. 2004 Jan-Feb;54(1):8-29. doi: 10.3322/canjclin.54.1.8. PMID 14974761
- [Background] Morson BC. Precancerous and early malignant lesions of the large intestine. Br J Surg. 1968 Oct;55(10):725-31. doi: 10.1002/bjs.1800551003. No abstract available. PMID 5681027
- [Background] Morson B. President's address. The polyp-cancer sequence in the large bowel. Proc R Soc Med. 1974 Jun;67(6 Pt 1):451-7. doi: 10.1177/00359157740676P115. No abstract available. PMID 4853754
- [Background] Cappell MS, Forde KA. Spatial clustering of multiple hyperplastic, adenomatous, and malignant colonic polyps in individual patients. Dis Colon Rectum. 1989 Aug;32(8):641-52. doi: 10.1007/BF02555767. PMID 2752850
- [Background] Rex DK, Chadalawada V, Helper DJ. Wide angle colonoscopy with a prototype instrument: impact on miss rates and efficiency as determined by back-to-back colonoscopies. Am J Gastroenterol. 2003 Sep;98(9):2000-5. doi: 10.1111/j.1572-0241.2003.07662.x. PMID 14499778
- [Background] Muto M, Katada C, Sano Y, Yoshida S. Narrow band imaging: a new diagnostic approach to visualize angiogenesis in superficial neoplasia. Clin Gastroenterol Hepatol. 2005 Jul;3(7 Suppl 1):S16-20. doi: 10.1016/s1542-3565(05)00262-4. PMID 16012987
- [Background] Kara MA, Peters FP, Rosmolen WD, Krishnadath KK, ten Kate FJ, Fockens P, Bergman JJ. High-resolution endoscopy plus chromoendoscopy or narrow-band imaging in Barrett's esophagus: a prospective randomized crossover study. Endoscopy. 2005 Oct;37(10):929-36. doi: 10.1055/s-2005-870433. PMID 16189764
- [Derived] Gross SA, Buchner AM, Crook JE, Cangemi JR, Picco MF, Wolfsen HC, DeVault KR, Loeb DS, Raimondo M, Woodward TA, Wallace MB. A comparison of high definition-image enhanced colonoscopy and standard white-light colonoscopy for colorectal polyp detection. Endoscopy. 2011 Dec;43(12):1045-51. doi: 10.1055/s-0030-1256894. Epub 2011 Oct 4. PMID 21971929